CLINICAL TRIAL: NCT01032265
Title: Web-based Management of Female Stress Urinary Incontinence. Evaluation of a Treatment Programme With Pelvic Floor Muscle Training and Elements of Cognitive Behavioural Therapy
Brief Title: Web-based Management of Female Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Swedish Council for Working Life and Social Research (Other); Jämtland County Council, Sweden (Other Government); Västernorrland County Council, Sweden (Other Government)
Responsible Party: Principal Investigator, Eva Samuelsson, Associate professor, Umeå University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAS dnr 2008-0952; VLL 759-2008 (Other: Umeå University and County Councils of Northern Sweden); VLL-68711 (Other: Umeå University and County Councils of Northern Sweden); SLS 2008-21468 (Other: Swedish Society of Medicine); Visare Norr Project nr 40/2009 (Other: County Councils of Northern Sweden); JLL LS/1073/2008 (Other: County Council of Jämtland); LVN 8160 (Other: County Council of Västernorrland)
Record Dates: First submitted 2009-12-12; First posted 2009-12-15 (Estimated); Results first posted 2013-03-13 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Female Stress Urinary Incontinence
Keywords: female; stress urinary incontinence; treatment; pelvic floor muscle training; cognitive behavioral therapy; internet; life style; pamphlet; eHealth
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Web-based treatment (Active Comparator): Web-based treatment with information (including life style), PFMT, elements of CBT and regular mail contact with an urotherapist
  Interventions: Behavioral: Web-based treatment with PFMT and elements of CBT
- Pamphlet treatment (Active Comparator): Information (including life style), and PFMT exercises.
  Interventions: Behavioral: Pamphlet treatment

INTERVENTIONS:
Behavioral: Web-based treatment with PFMT and elements of CBT — 125 women with stress urinary incontinence(SUI) participate in web-based treatment for 3 months. Treatment consists of information, PFMT and uses elements of CBT. It includes regular email contact with urotherapist.
  Arms: Web-based treatment
Behavioral: Pamphlet treatment — 125 women with SUI receive a pamphlet with information and a programme for PFMT.
  Arms: Pamphlet treatment

SUMMARY:
The purpose of this study is to determine whether treatment of female stress urinary incontinence using a web-based programme is effective.

DETAILED DESCRIPTION:
Female urinary incontinence is very common and affects up to one fourth of grownup women. It may reduce quality of life for those affected and costs for society are high. The most common type of urinary incontinence is stress urinary incontinence (SUI), i.e leakage when coughing, sneezing or jumping. There is no association between SUI and serious medical conditions. Thus investigation can be kept to a minimum, including structured history taking and a bladder diary for correct diagnosis. Treatment with lifestyle intervention and pelvic floor muscle training (PFMT) give improvement or cure in 60-70% of women. A small study indicates that treatment with cognitive behavioural therapy (CBT) may improve incontinence-related quality of life and symptoms of urinary incontinence. Web-based management of SUI has as far as we know never been evaluated in a randomized controlled study. The aim of this study is to determine if web-based management of female SUI, with a treatment using PFMT and elements of CBT is effective compared to treatment supported by a pamphlet. The duration of the treatment programme is three months, follow-up at four months, 1 year and two years.

ELIGIBILITY:
Inclusion Criteria:

* stress urinary incontinence
* leakage once a week or more often
* ability to read and write Swedish
* asset to computer with Internet connection

Exclusion Criteria:

* pregnancy
* former incontinence surgery
* known malignancy in lower abdomen
* difficulties with passing urine
* visual blood in urine
* intermenstrual bleeding
* severe psychiatric diagnosis
* neurological disease with affection on sensibility in legs or lower abdomen

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2009-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Samuelsson, MD, PhD, Study Chair — Department of Public Health and Clinical Medicine, Umeå University; Eva Samuelsson, MD, PhD, Principal Investigator — Department of Public Health and Clinical Medicine, Umeå University; Göran Umefjord, MD, PhD, Principal Investigator — Department of Public Health and Clinical Medicine, Umeå University
Locations (1):
- Umea University, Umeå, Sweden

REFERENCES:
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322
- [Derived] Sjostrom M, Umefjord G, Stenlund H, Carlbring P, Andersson G, Samuelsson E. Internet-based treatment of stress urinary incontinence: a randomised controlled study with focus on pelvic floor muscle training. BJU Int. 2013 Aug;112(3):362-72. doi: 10.1111/j.1464-410X.2012.11713.x. Epub 2013 Jan 25. PMID 23350826
- [Derived] Sjostrom M, Stenlund H, Johansson S, Umefjord G, Samuelsson E. Stress urinary incontinence and quality of life: a reliability study of a condition-specific instrument in paper and web-based versions. Neurourol Urodyn. 2012 Nov;31(8):1242-6. doi: 10.1002/nau.22240. Epub 2012 Apr 19. PMID 22517196
- See also: Click here for more information on this study. Web-based management of female stress urinary incontinence. Evaluation of a treatment programme using pelvic floor muscle training and elements of cognitive behavioural therapy. — http://www.econtinence.se

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Online recruitment via the project´s open access website, Dec 2009 - Oct 2010. Interested women answered an online survey for screening of the eligibility criteria. If eligible they were sent a postal questionnaire, including a 2-day bladder diary. Finally, to confirm the clinical diagnosis all women were interviewed by telephone by a urotherapist.
Pre-assignment Details: Randomisation was through a pre-specified computer-generated list, in blocks of eight. An independent administrator kept the list and consecutively allocated eligible participants to one of the two intervention groups. There was no blinding of group allocation to study participants, health care providers, or researchers.
Groups:
- Postal Treatment: Information (including life style), and PFMT exercises.
- Internet-based Treatment: Internet-based treatment with information (including life style), PFMT, elements of CBT and regular mail contact with an urotherapist
Period: Overall Study
Arm/Group | Postal Treatment | Internet-based Treatment
Started | 126 | 124
Completed | 113 | 107
Not Completed | 13 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Postal Treatment | Internet-based Treatment | Total
Number analyzed (Participants) | 126 | 124 | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (9.8) | 47.9 (10.6) | 48.6 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 124 | 250
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 126 | 124 | 250
Body Mass index [Mean (Standard Deviation); unit: kg/m2] | 24.5 (3.6) | 24.7 (4.2) | 24.6 (3.9)
Smoking [Number; unit: Participants]
  Smoker | 5 | 4 | 9
  Non-smoker | 121 | 120 | 241
Education [Number; unit: Participants]
  >=3 years at university level | 72 | 63 | 135
  < 3 years at university level | 28 | 25 | 53
  Lower | 26 | 36 | 62
Number of births (Parity) [Number; unit: Participants] — number of births
  Participants
    No childbirth | 7 | 11 | 18
    1 child | 15 | 20 | 35
    2 children | 62 | 61 | 123
    3 children | 31 | 21 | 52
    4 children | 11 | 11 | 22
Menopausal status [Number; unit: Participants]
  Postmenopausal | 48 | 43 | 91
  Not postmenopausal | 73 | 77 | 150
  Unknown | 5 | 4 | 9
Baseline characteristics for postal treatment group, internet-based treatment group and total [Number; unit: participants] | 126 | 124 | 250

OUTCOME MEASURES:

1. Primary Outcome: International Consultation on Incontinence Modular Questionnaire Urinary Incontinence Short Form (ICIQ-UI SF)
Description: summed symptom-score, range 0-21, with higher scores indicating greater severity.
Time Frame: baseline, 4 months
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Postal Treatment | Internet-based Treatment
Number analyzed (Participants) | 113 | 107
units on a scale
  Baseline | 10.3 (3.5) | 10.4 (3.1)
  4 month follow-up | 7.3 (3.9) | 6.9 (3.1)
Statistical Analysis 1: Comparison: Postal Treatment vs Internet-based Treatment; analysis between groups; Test type: Superiority or Other; p = 0.27, Mixed Models Analysis

2. Primary Outcome: International Consultation on Incontinence Modular Questionnaire Lower Urinary Tract Symptoms Quality of Life (ICIQ-LUTSqol)
Description: condition-specific quality of life, summed score, range 19-76, higher scores indicate greater impact on quality of life.
Time Frame: baseline, 4 months
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Postal Treatment | Internet-based Treatment
Number analyzed (Participants) | 113 | 107
units on a scale
  Baseline | 33.6 (8.2) | 33.6 (6.8)
  4 month follow-up | 28.8 (7.3) | 27.8 (6.0)
Statistical Analysis 1: Comparison: Postal Treatment vs Internet-based Treatment; analysis between groups; Test type: Superiority or Other; p = 0.52, Mixed Models Analysis

3. Secondary Outcome: EuroQol Five Dimensions Visual Analogue Scale (EQ5D-VAS)
Description: health-specific quality of life, range 0-100, higher scores indicate better quality of life.
Time Frame: baseline, 4 months
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Postal Treatment | Internet-based Treatment
Number analyzed (Participants) | 113 | 107
units on a scale
  Baseline | 79.2 (14.0) | 79.1 (13.6)
  4 month follow-up | 81.8 (13.9) | 83.3 (10.3)
Statistical Analysis 1: Comparison: Postal Treatment vs Internet-based Treatment; analysis between groups; Test type: Superiority or Other; p = 0.30, Mixed Models Analysis

4. Secondary Outcome: Usage of Incontinence Aids
Description: Only those using incontinence aids at baseline were included in the analysis.
Time Frame: baseline, 4 months
Population: Intention-to-treat
Measure: Number; unit: participants
Arm/Group | Postal Treatment | Internet-based Treatment
Number analyzed (Participants) | 82 | 79
participants
  No use | 11 | 17
  Less than before | 23 | 30
  Same as before | 46 | 32
  More than before | 2 | 0
Statistical Analysis 1: Comparison: Postal Treatment vs Internet-based Treatment; analysis between groups; Test type: Superiority or Other; p = 0.02, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Patient Satisfaction
Time Frame: 4 months
Population: Intention-to-treat
Measure: Number; unit: participants
Arm/Group | Postal Treatment | Internet-based Treatment
Number analyzed (Participants) | 113 | 107
participants
  very good | 15 | 46
  good | 56 | 43
  neither good or bad | 31 | 13
  bad | 8 | 3
  very bad | 3 | 0
  Missing | 0 | 2
Statistical Analysis 1: Comparison: Postal Treatment vs Internet-based Treatment; analysis between groups; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Incontinence Episode Frequency (IEF)
Description: number of incontinence episodes per week
Time Frame: baseline, 4 months
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: episodes per week
Arm/Group | Postal Treatment | Internet-based Treatment
Number analyzed (Participants) | 113 | 107
episodes per week
  Baseline | 9.4 (8.6) | 12.7 (12.0)
  4 month follow-up | 4.4 (6.7) | 4.8 (7.7)
Statistical Analysis 1: Comparison: Postal Treatment vs Internet-based Treatment; analysis between groups; Test type: Superiority or Other; p = 0.23, negative binomial regression

7. Secondary Outcome: Patient's Global Impression of Improvement Scale (PGI-I)
Time Frame: 4 months
Population: Intention-to-treat
Measure: Number; unit: participants
Arm/Group | Postal Treatment | Internet-based Treatment
Number analyzed (Participants) | 113 | 107
participants
  very much better | 4 | 12
  much better | 26 | 31
  a little better | 60 | 48
  no change | 19 | 13
  a little worse | 3 | 1
  much worse | 1 | 0
  very much worse | 0 | 0
  Missing | 0 | 2
Statistical Analysis 1: Comparison: Postal Treatment vs Internet-based Treatment; analysis between groups; Test type: Superiority or Other; p = 0.01, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Postal Treatment | Internet-based Treatment
Serious Adverse Events (participants affected / at risk) | 0/126 | 0/124
Other Adverse Events (participants affected / at risk) | 0/126 | 1/124
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Postal Treatment (N=126) | Internet-based Treatment (N=124)
Lower abdominal pain when performing pelvic floor muscle training (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No